CLINICAL TRIAL: NCT06889246
Title: Open-label, Single-center Clinical Trial to Evaluate the Anti-gastroesophageal Reflux Effect of Anvitra Gastric Suspension Health Supplements on Outpatients With Gastroesophageal Reflux at Hai Phong Medical University Hospital in 2024
Brief Title: The Anti-gastroesophageal Reflux Effect of Anvitra Gastric Suspension on Outpatients With Gastroesophageal Reflux Disease
Acronym: ANVITRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haiphong University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HPMU.CTBE/P0324; 02/2024/HD/AV-YDHP (Other Grant/Funding Number: Anvy Joint Stock Company)
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: GERD (Heartburn, Regurgitation, and Dyspepsia) Frequency; GERD (Heartburn, Regurgitation, and Dyspepsia) Severity
Keywords: Anvitra Gastric Suspension; GERD treatment; heartburn relief; regurgitation relief; dyspepsia relief
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Dyspepsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anvitra Gastric Suspension (Experimental): This arm includes 24 patients who receive the health supplement Anvitra Gastric Suspension. Participants take the product orally, 1 packet per dose, 30 minutes after breakfast, lunch and dinner, for 14 days.
  Interventions: Dietary Supplement: Anvitra Gastric Suspension

INTERVENTIONS:
Dietary Supplement: Anvitra Gastric Suspension — Anvitra Gastric Suspension is provided as a liquid oral preparation, designed with a pleasant flavor to ensure compliance in patients. The intervention involves administering 1 packet (15 ml) per dose three times daily, taken orally 30 minutes after meals, for a duration of 14 days. The supplement is intended to alleviate symptoms of GERD (heartburn, regurgitation, and dyspepsia). Anvitra Gastric Suspension has been widely used in clinical and community settings, with a favorable safety profile and reported effectiveness in GERD treament.

SUMMARY:
This is an open-label, single-center clinical trial evaluating the efficacy and safety of Anvitra Gastric Suspension health supplements in adult patients with gastroesophageal reflux. Participants will be given Anvitra for 14 consecutive days and will continue to be monitored for 7 days after the intervention. The study aims to assess improvements in GERD (gastroesophageal reflux disease) symtoms, as well as monitor adverse events associated with the interventions. Data will be collected over a 22-day period, including screening, treatment, and follow-up phases.

DETAILED DESCRIPTION:
The study spans 22 days for each participant, consisting of three phases:

1. Screening Phase (1 day): Eligibility determined based on inclusion and exclusion criteria.
2. Treatment Phase (14 days): Daily administration of the research product.
3. Follow-Up Phase (7 days): Monitoring of post-treatment outcomes.

Visit 1 After clinical examination, patients who meet the criteria for participation in the study, with a preliminary diagnosis of gastroesophageal reflux, the participant signs the consent form, the participant is checked for vital signs, paraclinical tests, clinical examination, and answers to the reflux disease questionnaire (RDQ). The study accepts the results of previous esophagogastric endoscopy within 28 days. The results of the endoscopy will be used to exclude other diseases of the digestive tract according to the exclusion criteria. The participant will be instructed to stop all drugs or any products that have the effect of reducing gastric acid secretion, anti-reflux and drugs that can aggravate reflux. At the end of Visit 1, participants will be provided with Anvitra Gastric Suspension for approximately 14 days until Visit 2. Participants will be instructed and self-administered Anvitra Gastric Suspension for the first time under the supervision of study site staff at Visit 1.

The investigator will contact daily to check the product usage history, remind participants to use the product and record any AEs/SAEs by using RDQ to assess the change in severity of symptoms each day.

Visit 2 On the morning of Day D15, all participants must carefully record the time of the last study intervention (evening of Day D14). Participants will be checked for vital signs, paraclinical tests, clinical examination, and answer the RDQ.

A telephone follow-up will occur approximately 7 days after (day D21) the last treatment dose to continue recording of AEs/SAEs.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older at the time of signing the ICF
2. Diagnosis of GERD
3. Los Angeles Grade A or B esophagitis
4. Symptoms of heartburn, reflux, or dyspepsia
5. The participant is willing and able, in the opinion of the investigator, to modify current GERD therapy as required by the protocol.
6. Ability to sign an informed consent form for participation in the study as described in Appendix A, including compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

1. Concomitant esophageal stenosis, tumors, esophageal cancer, Barrett's esophagus, stomach cancer, gastric ulcer: confirmed by the results of esophagogastroduodenoscopy at the first examination and/or medical records
2. History of other gastrointestinal diseases, severe diseases of other organs
3. Esophagitis grade C, D according to the Los Angeles classification
4. Unable to perform esophagogastroduodenoscopy: esophageal diseases that can cause esophageal perforation (esophageal burns due to chemicals, drugs causing esophageal stenosis), thoracic aortic aneurysm, heart failure, myocardial infarction, hypertensive crisis, respiratory failure, difficulty breathing due to any cause, severe cough, severe scoliosis, elderly patients, mentally ill patients who cannot cooperate, hypotension, patients who do not agree to perform. 5. Severe hepatic or renal impairment and other chronic medical conditions.

6. Current use of medications that affect the gastrointestinal tract, medications that are known to cause or aggravate gastroesophageal reflux disease.

7. Participation in another clinical study with a study intervention performed within the last 14 days.

8. Planned hospitalization during the study.

9. The investigator's judgment that the participant should not participate in the study if the participant is unable to comply with the study procedures, restrictions and requirements.

10. Women only: currently pregnant (confirmed by a positive pregnancy test), breastfeeding or planning to become pregnant during the study, or not using acceptable contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
GERD Condition Improvement Assessment | Day 15 and Day 21
  Assessment of changes in GERD (heartburn, regurgitation, and dyspepsia) severity and frequency using the Reflux Disease Questionnaire (RDQ). The RDQ uses a scale ranging from 0 (Not at all) to 5 (Extremely severe). Higher scores indicate worse outcomes.

SECONDARY OUTCOMES:
Adverse Events Monitoring | Throughout the 21-Day Study Period
  Monitoring and recording of adverse events associated with Anvitra Gastric Suspension throughout the study period

CONTACTS AND LOCATIONS:
Locations (2):
- Vietnam (2):
  - Center for Clinical Trial and Bioequivalence Study, Haiphong, Hải Phòng
  - Center for Clinical Trial and Bioequivalence Study, Haiphong University of Medicine and Pharmacy, Haiphong

IPD SHARING:
Plan to Share IPD: No
As the request of the sponsor